CLINICAL TRIAL: NCT04886414
Title: Implementation and Evaluation of Home-based Care and Hand Hygiene Interventions in Honduras
Brief Title: Home-based Care and Hand Hygiene Interventions in Honduras
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); Ministry of Health, Honduras (Other Government)
Responsible Party: Principal Investigator, Eric J. Nilles, M.D.,M.S.C., Assistant Professor, Brigham and Women's Hospital
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: 2021P001143
Record Dates: First submitted 2021-05-10; First posted 2021-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Covid19
Keywords: Home-Based Care; Water, Sanitation and Hygiene; Alcohol-Based Hand Sanitizer; Triage; Post-Covid Syndrome; Community Health Workers
MeSH Terms: conditions — COVID-19 | interventions — Ethanol

STUDY DESIGN:
Intervention Model Description: Participants will be block randomized to one of four possible home-based care strategies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Phone-based monitoring without blood oxygenation monitoring with ABHS (Experimental): Study staff will perform daily phone-based assessments using standardized electronic study tools (tablets). Clinical features will be documented on a phone-based patient monitoring form. Subjects will received a home-based care kit that contains alcohol-based hand sanitizer (ABHS).
  Interventions: Other: Phone-based monitoring; Other: Alcohol-based hand sanitizer
- Phone-based monitoring without blood oxygenation monitoring without ABHS (Experimental): Study staff will perform daily phone-based assessments using standardized electronic study tools (tablets). Clinical features will be documented on a phone-based patient monitoring form. Subjects will received a home-based care kit that does not contain alcohol-based hand sanitizer.
  Interventions: Other: Phone-based monitoring
- Phone-based monitoring with blood oxygenation monitoring with ABHS (Experimental): Study staff will perform daily phone-based assessments using standardized electronic study tools (tablets). Clinical features and oxygen saturation levels will be documented on a phone-based patient monitoring form. Oxygen saturation level will be assessed four times per day (morning, midday, evening, plus during the phone-based assessment) by the patient and/or family member and the lowest stable (i.e. without substantial fluctuations) level recorded during a monitoring period of one minute will be recorded and registered. Patient's will be provided monitoring sheets to record the times and dates of the oxygen saturation levels. Subjects will received a home-based care kit that contains alcohol-based hand sanitizer.
  Interventions: Other: Phone-based monitoring; Other: Oxygen saturation monitoring; Other: Alcohol-based hand sanitizer
- Phone-based monitoring with blood oxygenation monitoring without ABHS (Experimental): Study staff will perform daily phone-based assessments using standardized electronic study tools (tablets). Clinical features and oxygen saturation levels will be documented on a phone-based patient monitoring form. Oxygen saturation level will be assessed four times per day (morning, midday, evening, plus during the phone-based assessment) by the patient and/or family member and the lowest stable (i.e. without substantial fluctuations) level recorded during a monitoring period of one minute will be recorded and registered. Patient's will be provided monitoring sheets to record the times and dates of the oxygen saturation levels. Subjects will received a home-based care kit that does not contain alcohol-based hand sanitizer.
  Interventions: Other: Phone-based monitoring; Other: Oxygen saturation monitoring

INTERVENTIONS:
Other: Phone-based monitoring — Study staff will perform daily phone-based assessments using standardized electronic study tools (tablets). Clinical features will be documented on a phone-based patient monitoring form.
Other: Oxygen saturation monitoring — Oxygen saturation will be monitored and recorded at regular intervals.
  Arms: Phone-based monitoring with blood oxygenation monitoring with ABHS; Phone-based monitoring with blood oxygenation monitoring without ABHS
Other: Alcohol-based hand sanitizer — Alcohol-based hand sanitizer will be distributed to subjects.
  Arms: Phone-based monitoring with blood oxygenation monitoring with ABHS; Phone-based monitoring without blood oxygenation monitoring with ABHS

SUMMARY:
This study aims to enroll patients with acute infection with Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) who do not meet criteria for hospital admission according to protocols developed by the Honduras Ministry of Health (MOH). Patients who are triaged to home must also be over the age of 60 years or have one high risk comorbidity and be over 45 years in order to meet inclusion criteria. These patients will be randomly assigned to one of four home-based care strategies, which may or may not include regular blood oxygenation monitoring and provision of alcohol-based hand-rub. Patients will be followed until resolution of their acute illness, and data will be collected on feasibility, impact and acceptance of the intervention. Some patients will be followed for up to one year to monitor for post-Coronavirus Disease 2019 (COVID-19) symptoms.

DETAILED DESCRIPTION:
Rationale:

This project is intended to enhance the existing MOH home-based care approach by providing additional resources and monitoring for patients with COVID-19 that are triaged to Home-based care (HBC) by MOH triage clinicians. In addition, given limited data on which home-based care strategies most effectively and efficiently minimize poor outcomes, we aim to monitor four discrete home-based care approaches. Assignment to home-based care approach will be randomized. Given the primary goal of the project is to reduce morbidity and mortality due to the COVID-19 pandemic, we will not include a control arm.

Setting:

The project location will be the designated municipalities in Honduras. Activities will be conducted in the existing MOH triage (known by the Spanish acronym for Temporary Triage and Stabilization Centers: "CETTE's") and other health centers. Selection of target centers will be performed in collaboration with the Honduras MOH and based on criteria including current and projected COVID-19 hotspots, mortality data and logistical considerations including access and security.

Project Population:

The study population is patients ≥ 45 years old with COVID-19 assessed to be higher-risk for potentially poor outcomes but defined in the triage center as clinically stable and suitable for home-based care according to existing Honduras MOH COVID-19 protocols. The assessment of which patients will be discharged to home will be conducted by MOH clinicians according to existing MOH protocols. Patients suspected of having COVID-19 will have the infection confirmed by rapid antigen test prior to enrollment.

Inclusion criteria:

* Patients presenting to triage centers with suspected acute infection with SARS-CoV-2.
* Positive rapid antigen test for SARS-CoV-2
* Patients triaged to HBC by MOH clinicians according to existing MOH policies and protocols.
* Greater than 60 years of age OR greater than 45 years of age AND at least one comorbidity which increases risk for poor outcomes due to COVID-19.
* Live or work in the city where the study is being implemented
* Agrees to participate and signs informed consent

Exclusion criteria:

* Less than 45 years of age
* Incapable of giving assent to participate due to medical condition at the time of enrollment

Recruitment procedures:

Screening and recruitment will occur in the health facility or CETTE. Patients that are evaluated by MOH clinicians and triaged to HBC will undergo further screening by project staff to assess if they meet project inclusion criteria. Those that (i) are triaged to HBC by MOH clinicians and (ii) meet the additional project inclusion criteria will be enrolled by study staff.

Home based care strategies

Participants will be assigned at the time of enrollment to one of two following home-based care strategies using a block randomization approach:

* Strategy 1: Study staff will perform daily phone-based assessments using standardized electronic study tools (tablets). Clinical features will be documented on a phone-based patient monitoring form.
* Strategy 2: Study staff will perform daily phone-based assessments using standardized electronic study tools (tablets). Clinical features and oxygen saturation levels will be documented on a phone-based patient monitoring form. Oxygen saturation level will be assessed three times per day (morning, evening, plus during the phone-based assessment) by the patient and/or family member and the lowest stable (i.e. without substantial fluctuations) level recorded during a monitoring period of one minute will be recorded and registered. Patient's will be provided monitoring sheets to record the times and dates of the oxygen saturation levels.

Referral to higher level of care:

Patients meeting referral criteria of oxygen saturation (SpO2)<92% or other alarm signs will be referred to the nearest CETTE or hospital care according to existing MOH guidelines.

Home-based care kits and strategies:

All study participants will receive COVID-19 HBC kits that will include soap, face masks, information sheets on COVID-19 prevention, and other supplies. Half the COVID-19 home kits will include ABHS. Patients will be assigned to study strategies based on they day they present to the CETTE, with the four strategies rotating in order. Patients assigned to Strategy 2 will be supplied with a portable pulse oximeter and trained on use and measurement by study staff prior to discharge from the triage center. Patients who are triaged to HBC by CETTE's but are deemed ineligible for study enrollment may also be provided with an HBC kit if resources are available.

Discharge from daily clinical monitoring:

All patients will receive daily monitoring until they are discharged from the daily monitoring program. Criteria for discharge are:

1. Ten days post-symptoms onset and 24 hours without fever. Patients meeting these criteria will be discharged from the daily monitoring program. If a patient continues to experience fever more than 10-days post-symptoms onset they will continue to receive daily monitoring until they are fever-free for more than 24 hours.
2. Hospitalization (over 24 in the hospital). If a patient is hospitalized they will be discharged from the daily monitoring program. Patients that are not hospitalized will continue in the daily monitoring program until criteria #1 is met.

Data collection and survey tools:

1. Baseline survey All enrolled patients will complete a baseline survey that will include demographic and clinical information, risk factors, hand hygiene practices and other WASH variables, and sociobehavioral questions. Survey questions will include timing and nature of symptoms, and COVID-19 compatible symptoms, if anyone else in the household has had COVID-19 symptoms in the past 30 days, and if so, when they began and how long they lasted. The enrollment survey will also assess risk factors of the participant and household members such as which household members leave the house for work or school and if there are any other possible exposures to COVID-19. Specific questions about the WASH component include assessing the participants' knowledge, attitudes, and practices about hand hygiene in the month prior to visiting the triage center. The enrollment survey will assess access to hand hygiene resources in the participants' homes by asking about access to water and soap in the participants' homes. The estimated time to complete baseline enrollment and questionnaire is 20-25 minutes.
2. Daily acute COVID-19 symptoms Study staff will document clinical features including vital signs and alarm signs or symptoms during each daily follow-up visit using a standardized form. Data on COVID-19 compatible symptoms among household members will also be collected; gender and age of household members will be recorded but no additional identifiable information will be collected. These questions will allow investigators to assess if other household members were infected or become infected with COVID-19 as a result of likely in-home transmission or community acquired infection. Daily clinical follow-up evaluations are estimated to take 10 minutes.
3. Inpatient chart review Patients with SpO2<92% or who otherwise are decompensating are referred back to the triage centers or to a higher level. In these cases, investigators will abstract data on clinical course and patient outcomes from relevant health facilities. A standard data abstraction form will be completed for study subjects who were hospitalized or received outpatient supplemental oxygen in the CETTE. Data collected will include patients' disposition at admission and discharge, treatment received, and length of stay. Each inpatient chart review is estimated to take two hours including travel time for study staff.
4. Follow-up hand hygiene assessment Serial follow-up WASH survey will be administered every week and at discharge (from acute COVID-19 daily monitoring) during the daily follow-up contacts for the HBC study. The follow-up survey will repeat questions about hand hygiene practices to assess changes in hand hygiene behavior after visiting the triage center and receiving the HBC kit. Last, the follow up survey will also assess the safe usage of the ABHS in the home by asking if there have been any adverse events (e.g. splash in eye or ingestion). This questionnaire is estimated to take 5 minutes.
5. Exit interview from acute COVID-19 monitoring All study participants will be administered a phone-based exit interview to understand their opinions and level of satisfaction with the care provided in each study arm. This questionnaire is estimated to take 5 minutes.
6. Assessment of study staff perceptions After finishing follow up for their tenth HBC patient, study staff will complete an electronic survey to assess staff acceptance and feasibility of HBC with or without pulse oximetry. This questionnaire is estimated to take 5 minutes.
7. Chronic COVID-19 symptoms Following discharge from acute COVID-19 daily monitoring, study staff will administer phone surveys to all study participants a minimum of every 3 months through the course of the project to assess COVID-19 sequelae and use of health services. Participants may be offered a medical assessment during the follow-up period of symptoms monitoring. Data will be collected using a standardized Post-Covid Conditions Questionnaire. Longitudinal follow-up phone surveys to assess for chronic COVID-19 symptoms are estimated to take 5 minutes.

Indicators:

Specific indicators will be used to assess the feasibility, impact and acceptance of the HBC intervention. Although final indicators may be updated and/or modified, the preliminary set of indicators are listed below.

1. Feasibility

   * Proportion that receive the prescribed follow-up plan
   * Proportion with complete pulse oximetry data, for relevant arms
   * Loss to follow-up
2. Referral to higher level of care

   * Proportion referred to higher level care due to hypoxia (i.e. SpO2 < 92%)
   * Proportion referred to higher level care due to alarm symptoms
   * Proportion referred to higher level care for any other reason
   * Proportion referred that reach higher level of care within 24 hours
   * Proportion who successfully complete HBC without requiring referral
   * Disposition after referral (home, admission, other)
   * SpO2 level upon arrival to higher level of care
   * Other clinical measures upon arrival to higher level of care
3. Impact on patient outcomes:

   * Duration of hospitalization (days)
   * Duration of ICU and/or ventilator requirement*
   * Mortality*
4. Acceptability

   * Perception of utility/benefit of strategy (study staff/patients/family)
   * Perception of ease of implementation of strategy (study staff)
   * Changes in hand hygiene behavior

ELIGIBILITY:
Inclusion criteria:

* Patients presenting with acute infection with SARS-CoV-2.
* Patients test positive for SARS-CoV-2 with rapid antigen test.
* Patients triaged to HBC by SESAL clinicians according to existing SESAL policies and protocols.
* Greater than 60 years of age OR greater than 45 years AND at least one comorbidity which increases risk for poor outcomes due to COVID-19.
* Live or work in the city where the study is being implemented
* Agrees to participate and signs informed consent

Exclusion criteria:

* Less than 45 years of age
* Incapable of giving assent to participate due to medical condition at the time of enrollment

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1821 (Actual)
Dates: Start 2022-03-31 (Actual); Primary Completion 2023-01-15 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Disposition after referral | 28 days
  Disposition (home, admission, other) for those referred to a higher level of care
Duration of hospitalization | 90 days
  Duration of hospitalization (days) for those who are admitted
Duration of ICU and/or ventilator requirement | 90 days
  Duration of ICU and/or ventilator requirement (days) for those requiring critical care
Mortality | 90 days
  Death prior to discharge from acute COVID-19 monitoring

OTHER OUTCOMES:
Proportion that receive the prescribed follow-up plan | 28 days
  Proportion that receive the prescribed home-based care follow-up plan
Proportion with complete pulse oximetry data | 28 days
  Proportion with complete pulse oximetry data, for relevant arms
Loss to follow-up | 90 days
  Loss to follow-up
Reason for referral | 28 days
  Proportion referred to higher level care due to hypoxia (i.e. SpO2 < 92%), due to alarm symptoms or for any other reason.
Proportion referred that reach higher level of care within 24 hours | 28 days
  Proportion referred that reach higher level of care within 24 hours
Proportion who successfully complete HBC without requiring referral | 28 days
  Proportion who successfully complete HBC without requiring referral
SpO2 level upon arrival to higher level of care | 28 days
  SpO2 (%) level upon arrival to higher level of care
Other clinical measures upon arrival to higher level of care | 28 days
  Other clinical measures (e.g. vital signs, alarm signs) upon arrival to higher level of care for those who are referred
Perception of utility/benefit of strategy (CHW/patients/family) | 28 days
  Perception of utility/benefit of strategy based on qualitative interviews with community health workers, patients and family
Perception of ease of implementation of strategy | 28 days
  Perception of ease of implementation of strategy based on interview with community health workers
Changes in hand hygiene behavior | 28 days
  Changes in hand hygiene behavior reported by participants

CONTACTS AND LOCATIONS:
Locations (1):
- COVID-19 Triage Centers, Tegucigalpa, Francisco Morazán Department, Honduras

REFERENCES:
- [Derived] Roberts KW, Alvarez B, de St Aubin M, Diaz O, Garnier S, Schnorr CD, Cruz S, Pavon L, Ochoa A, See R, Medice S, Santos HM, Ochoa J, Solis S, Dumas D, Baldwin M, Martinez A, Hakim A, Nilles E. Impact of self-administered pulse oximetry among non-hospitalized patients at risk of severe COVID-19 in Honduras: A pragmatic, cluster-randomized trial with temporal clustering. PLOS Glob Public Health. 2025 Nov 7;5(11):e0004618. doi: 10.1371/journal.pgph.0004618. eCollection 2025. PMID 41202024